CLINICAL TRIAL: NCT01254760
Title: Comparison of Two Multifocal Contact Lenses Worn on a Daily Disposable Basis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: P-416-C-001 Sub 04
Record Dates: First submitted 2010-12-03; First posted 2010-12-07 (Estimated); Results first posted 2012-02-17 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-01

CONDITIONS: Presbyopia; Myopia
MeSH Terms: conditions — Presbyopia; Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational multifocal / Commercial multifocal (Other): Investigational multifocal contact lenses worn first, with commercial multifocal contact lenses worn second. Each product worn bilaterally on a daily wear, daily disposable basis for 5 days.
  Interventions: Device: Nelfilcon A multifocal contact lens, investigational; Device: Nelfilcon A multifocal contact lens, commercial
- Commercial multifocal / Investigational multifocal (Other): Commercial multifocal contact lenses worn first, with investigational multifocal contact lenses worn second. Each product worn bilaterally on a daily wear, daily disposable basis for 5 days.
  Interventions: Device: Nelfilcon A multifocal contact lens, investigational; Device: Nelfilcon A multifocal contact lens, commercial

INTERVENTIONS:
Device: Nelfilcon A multifocal contact lens, investigational — Investigational, soft, multifocal contact lens for daily wear, daily disposable use.
Device: Nelfilcon A multifocal contact lens, commercial — Commercially marketed, soft, multifocal contact lens FDA-approved for daily wear, daily disposable use.
  Other Names: Focus® DAILIES® Progressive

SUMMARY:
The purpose of this trial is to evaluate and compare the clinical performance of two multifocal contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Age 41 to 68 (inclusive).
* Spectacle add between +0.75 and +2.75D (inclusive).
* Habitual spectacle prescription ≤ 1.00DC (cyl).
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Eye injury or surgery within twelve weeks of enrollment.
* Pre-existing ocular irritation that would preclude contact lens fitting.
* Currently enrolled in a clinical trial.
* Prior refractive surgery.
* Other protocol-defined exclusion criteria may apply.

Ages: 41 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2010-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 79 participants were recruited at 7 US sites from December 3, 2010, to January 20, 2011.
Pre-assignment Details: Seven participants were enrolled in the study but not dispensed due to failed inclusion/exclusion criteria (2); unsatisfactory vision (2); unacceptable comfort (1); and subject withdrawal (2). These participants are included in the Actual Enrollment calculation, but not Participant Flow or Baseline Characteristics calculations.
Period: First Period, 5 Days of Wear
Arm/Group | Investigational Multifocal / Commercial Multifocal | Commercial Multifocal / Investigational Multifocal
Started | 34 | 38
Completed | 34 | 38
Not Completed | 0 | 0
Period: Second Period, 5 Days of Wear
Arm/Group | Investigational Multifocal / Commercial Multifocal | Commercial Multifocal / Investigational Multifocal
Started | 34 | 38
Completed | 34 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: This reporting group includes all enrolled and dispensed participants.
Arm/Group | Overall
Number analyzed (Participants) | 72
Age Continuous [Mean (Standard Deviation); unit: years] | 50.1 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: End of Day Comfort
Description: End of day comfort was interpreted and reported by the participant on a questionnaire as a single, retrospective evaluation of 5 days of wear. End of day comfort was measured on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 5 days of wear, lenses replaced daily
Population: Analysis conducted per protocol, with exclusions due to reasons such as: major protocol deviations as determined by masked review; discontinuations; and/or missing responses.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Nelfilcon A Investigational: Nelfilcon A investigational contact lenses worn bilaterally on a daily wear, daily disposable basis for 5 days
- Nelfilcon A Commercial: Nelfilcon A commercial contact lenses worn bilaterally on a daily wear, daily disposable basis for 5 days
Arm/Group | Nelfilcon A Investigational | Nelfilcon A Commercial
Number analyzed (Participants) | 71 | 71
Units on a scale | 7.7 (2.2) | 7.2 (2.3)

2. Primary Outcome: End of Day Dryness
Description: End of day dryness was interpreted and reported by the participant on a questionnaire as a single, retrospective evaluation of 5 days of wear. End of day dryness was measured on a 10-point scale, with 1 being very dry and 10 being not dry.
Time Frame: 5 days of wear, lenses replaced daily
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Nelfilcon A Investigational | Nelfilcon A Commercial
Number analyzed (Participants) | 71 | 71
Units on a Scale | 7.2 (2.5) | 6.9 (2.5)

3. Primary Outcome: Handling at Removal
Description: Handling at removal was interpreted and reported by the participant on a questionnaire as a single, retrospective evaluation of 5 days of wear. Handling at removal was measured on a 10-point scale, with 1 being poor/difficult and 10 being excellent/easy.
Time Frame: 5 days of wear, lenses replaced daily
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Nelfilcon A Investigational | Nelfilcon A Commercial
Number analyzed (Participants) | 71 | 70
Units on a Scale | 8.7 (1.6) | 8.2 (2.1)

4. Primary Outcome: Overall Vision
Description: Overall vision was interpreted and reported by the participant on a questionnaire as a single, retrospective evaluation of 5 days of wear. Overall vision was measured on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 5 days of wear, lenses replaced daily
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Nelfilcon A Commercial: Nelfilcon A commercial contact lenses worn in bilaterally on a daily wear, daily disposable basis for 5 days
Arm/Group | Nelfilcon A Investigational | Nelfilcon A Commercial
Number analyzed (Participants) | 70 | 71
Units on a Scale | 7.2 (1.9) | 6.2 (2.1)

5. Secondary Outcome: Overall Fit
Description: Overall lens fit was assessed by the investigator at study visit using a biomicroscope, which magnifies the appearance of the contact lens on the participant's eye. Lens fit was assessed by eye and graded on a 5-point scale, with 2=unacceptably loose, 1= acceptably loose, 0=optimal, -1=acceptably tight, and -2=unacceptably tight
Time Frame: Day 5, lenses replaced daily
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: Eyes
Arm/Group | Nelfilcon A Investigational | Nelfilcon A Commercial
Number analyzed (Participants) | 69 | 69
Number analyzed (Eyes) | 138 | 138
Units on a Scale | 0.0 (0.5) | -0.1 (0.6)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the trial: 53 days
Description: This reporting group includes all enrolled and exposed participants.
Groups:
- Nelfilcon A Investigational: Nelfilcon A investigational contact lenses worn in both eyes on a daily wear, daily disposable basis for 5 days
- Nelfilcon A Commercial: Nelfilcon A commercial contact lenses worn in both eyes on a daily wear, daily disposable basis for 5 days
Arm/Group | Nelfilcon A Investigational | Nelfilcon A Commercial
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/77
Other Adverse Events (participants affected / at risk) | 0/77 | 0/77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.